CLINICAL TRIAL: NCT00001503
Title: Follow-up for Patients Previously Enrolled on the Center for Cancer Research Protocols
Brief Title: Follow-up Protocol for Patients With Cancer/AIDS/Skin Disease
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960071; 96-C-0071; NCT00296075 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Melanoma; Ovarian Cancer; Prostate Cancer; Breast Cancer; Lymphoma
Keywords: Cancer; Late-effects; Survival; Follow-Up; Natural History
MeSH Terms: conditions — Melanoma; Ovarian Neoplasms; Prostatic Neoplasms; Breast Neoplasms; Lymphoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/All Patients: Patients who were previously enrolled on a CCR protocol and need follow-up by CCR Investigators.

SUMMARY:
This protocol is to provide follow-up medical/surgical visits for DCS patients who are long term survivors and may not currently be a participant entered on an active research protocol. No investigational treatments or standard treatments will be administered on this protocol.

DETAILED DESCRIPTION:
Background:

* Patients enrolled on CCR clinical protocols may require long term follow-up to assess outcome (e.g., survival) or the effects of prior therapy.
* Keeping the primary treatment protocols open after accrual is complete in order to follow patients for long term outcome is an administrative burden on investigators and the IRB.

Objectives:

-To provide follow-up for patients who are long term survivors previously enrolled Center for Cancer Research (CCR) trial but who may not currently be enrolled on a research protocol.

Eligibility:

-Patients who were previously enrolled on a CCR protocol and who are not eligible for an active NCI intramural primary research protocol.

Design:

* The medical procedures/tests will be based on the patient's diagnosis, treatment and supporting clinical information. This is a follow-up study in which only standard tests and procedures are to be performed.
* Clinical information that is relevant to the patients prior protocols will be collected for research purposes.
* Procedures that entail more than minimal risk to the patient should not be performed for research purposes on this protocol.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Patients of any age who were previously enrolled on a CCR protocol.

Not eligible for or unwilling to participate in an active NCI intramural primary research protocol.

CCR investigator decides it is in the best interests of the patient and the CC for the patient to be seen in follow-up visits at the NIH.

Patient or Legally Authorized Representative (LAR)/guardian is able to provide informed consent.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of any age who were previously enrolled on a CCR protocol and need follow-up by CCR Investigators.
Sampling Method: Non-Probability Sample
Enrollment: 1031 (Actual)
Dates: Start 1996-09-19 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
To provide follow-up for patients who are long term survivors previously enrolled Center for Cancer Research (CCR) trial but who may not currently be enrolled on a research protocol | 30 years
  Provision of a mechanism to follow selected CCR patients when their protocols have been terminated.

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1996-C-0071.html